CLINICAL TRIAL: NCT03748498
Title: Effect of Low Level Laser Therapy on Postoperative Pain After Single Visit Endodontic Treatment
Brief Title: Effect of Low Level Laser Therapy on Post-endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Adem Günaydin, research assistant, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ag134134
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain
Keywords: laser; pulpitis; pain
MeSH Terms: conditions — Pain, Postoperative; Pulpitis; Pain | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized, placebo-controlled trial of 2 groups.
Who Masked: Investigator
Masking Description: All procedures were conducted by one clinician , and assignment was concealed from the clinician who performed the laser applications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser group (Experimental): Low level laser was applied for 60 second per tooth using Nd-YAG laser.
  Interventions: Device: laser
- placebo group (Placebo Comparator): The same procedures as in the laser group were performed, been completed but the laser was not activated in this group.
  Interventions: Device: laser

INTERVENTIONS:
Device: laser — Application of the laser was performed through root canal and to the buccal mucosa over the apices of the target tooth

SUMMARY:
This study was designed as a randomized, placebo-controlled trial of 2 groups. The treatment procedures were performed by one operator. After local anesthesia and rubber dam isolation, access cavity preparation was performed by diamond burs with high-speed hand pieces under the water cooling. . Instrumentation of procedures was performed by Reciproc R50 files. Irrigation protocol was completed, canal were dried, filled with gutta-percha cones and AH Plus sealer. After chemo- mechanical instrumentation and root canal filling procedures, LLLT was applied for 60 second per tooth using Nd-YAG laser ( λ=1064 nm,100 mJ, 10 Hz, 1-W) The same procedures as in the laser group were performed, been completed but the laser was not activated in this group. These patients were assigned as placebo group. Postoperative pain was measured and documented via the Visual Analogue Scale. Chi-square test was performed in analysis of the nominal data.There was statistically significant difference between groups at the 12th and 24th hours (p<.05). ). However, no statistically significant difference was found between the groups at the 4th, 8th, 48th, and 72th hours (p>.05). No statistically significant differences were detected between the groups in terms of demographic data (age and tooth number) except for gender (P > .05).LLLT can decrease postoperative pain after root canal treatment of single rooted teeth.

DETAILED DESCRIPTION:
The study was approved by the local ethics committee ....................., and informed consent was received from all participants. Study subjects were selected among patients who presented to the Department of Endodontics, Faculty of Dentistry ........................from September 2017 to March 2018.

Root canal treatment was planned for patients who participated in this study and have single root and single canal. Patients aged between 15 to 45 years. Exclusion criteria related with teeth were swelling or sinus tract, acute pain, periodontal probing greater than 3mm, internal and external resorption, fractured and cracked tooth, percussion sensitivity, and periapical index classification 3, 4, 5 according to Orstavik et al. (1986). Exclusion criteria related with systemic health of patients included diabetes, hypertension and cardiovascular pathologies, the use of analgesics and / or antibiotics at least one week before treatment, and using antidepressant drugs.The treatment procedures were performed by one operator (G.A.). Initially, patients' age, gender, and tooth number were recorded by the operator. 1.5 mL 2% articaine with 0.012 mg epinephrine (Ultracaine DS Forte; Aventis, Istanbul, Turkey) was used as local anesthetic. After rubber dam isolation, access cavity preparation was performed by diamond burs (ADIA Dental Burs, Turkey) with high-speed hand pieces under the water cooling. A #10 K- type (Kerr Corporation, Orange, CA) file was inserted to root canal to determine working length using an apex locator (Raypex, VDW). Working length was set as 1 mm shorter than the apical foramen and confirmed with periapical radiographs. Instrumentation of procedures was performed by Reciproc R50 files (VDW, Munich, Germany). Irrigation protocol was completed 5 mL 17% EDTA (Werax, Turkey) and 15 mL 2.5% sodium hypochlorite (NaOCl)(Wizard, Turkey ) with a side-vented needle (NaviTip needle; Ultradent Products Inc, South Jordan, UT). Subsequently, canal were dried with paper points and filled with gutta-percha cones and AH Plus sealer (Dentsply Maillefer). Lateral cold condensation technique was used for obturation. Finally, coronal access cavity was restored with a temporary restorative material (Cavit G; 3M ESPE, St Paul, MN). Permanent restoration was completed after the end of the experiment.A randomization was produced using through a website (http://www.random.org), after the clinician (G.A.) was completed all treatment procedures. All procedures were conducted by one clinician (C.E.B.), and assignment was concealed from the clinician who performed the laser applications (U.B.). Data analysis and interpretation were completed by the other researcher (C.F.) After chemo- mechanical instrumentation and root canal filling procedures, LLLT was applied for 60 second per tooth using Nd-YAG laser ( λ=1064 nm,100 mJ, 10 Hz, 1-W[Deka smart file, DEKA, Italy]). Application of the laser was performed through root canal and to the buccal mucosa over the apices of the target tooth. An application biostimulation tip was used to ensure a constant distance of 10 mm to the tissue.The same procedures as in the laser group were performed, been completed but the laser was not activated in this group. These patients were assigned as placebo group.Postoperative pain was measured and documented via the Visual Analogue Scale (VAS). VAS consists of a 100 mm line which is represented at one end by a sign 'No pain' and at the other end 'unbearable pain'. This form was given to the each patient and they were instructed to mark according to the pain intensity at 4th, 8th, 12th, 24th, 48th and 72th hours.There was statistically significant difference between groups at the 12th and 24th hours (p<.05). However, no statistically significant difference was found between the groups at the 4th, 8th, 48th, and 72th hours (p>.05). Aside from sex, No statistically significant differences were detected between the groups in terms of demographic data (age and tooth number) except for gender (P > .05). During in this study, no patient reported swelling, sinus tract, palpation pain and didn't need analgesics both in groups.Within the limitations of the present study, LLLT can decrease postoperative pain after root canal treatment of single rooted teeth.

ELIGIBILITY:
Inclusion Criteria:

* Root canal treatment was planned for patients who participated in this study and have single root and single canal. Patients aged between 15 to 45 years

Exclusion Criteria:

* Exclusion criteria related with teeth were swelling or sinus tract, acute pain, periodontal probing greater than 3mm, internal and external resorption, fractured and cracked tooth, percussion sensitivity, and periapical index classification 3, 4, 5 according to Orstavik et al. (1986).
* Exclusion criteria related with systemic health of patients included diabetes, hypertension and cardiovascular pathologies, the use of analgesics and / or antibiotics at least one week before treatment, and using antidepressant drugs.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation | 3 day
  Postoperative pain was measured and documented via the Visual Analogue Scale (VAS). VAS consists of a 100 mm line which is represented at one end by a sign 'No pain' and at the other end 'unbearable pain'.

CONTACTS AND LOCATIONS:
Overall Officials: ELİF BAHAR ÇAKICI, ASST. PROF., Principal Investigator — Ordu University
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided